CLINICAL TRIAL: NCT03716895
Title: Identifying Risk Factors for Complications in Severe Septic Shock
Brief Title: Severe Septic Shock Complications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Marc Vives, Clinical Research Lead. Department of Anesthesiology & Critical Care, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Other Study IDs: SSS-500
Record Dates: First submitted 2018-10-13; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Septic Shock
Keywords: Severe Septic Shock; Lactate clearance; Acute Kidney Injury; Days alive and free; Ventilation-free days; Vasopressor-free days
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adults older than 18 years old, admitted to the ICU with a Severe Septic Shock, requiring Norepinephrine at more than 0.25mcg/kg/min, who have signed informed consent form, will be consecutively included, from december 2018 to december 2019.

The primary goal is to look for risk factors associated with an increased in lactate clearance

Secondary goals are the following:

1. To look for risk factors associated with an increase risk of Hospital and ICU length of stay.
2. To look for risk factors associated with an increase risk of Acute Kidney Injury.
3. To look for risk factors associated with a decrease in days alive and free of Mechanical Ventilation, Vasopressors and Renal Replacement Therapy.
4. To look for risk factors associated with a decrease in Ventilator-free days.
5. To look for risk factors associated with a decrease in Vasopressor-free days.
6. To look for risk factors associated with an increase risk of in-hospital mortality.
7. To look for risk factors associated with an increase risk of Myocardial Infarction and myocardial injury.
8. To look for risk factors associated with an increase risk of Acute Respiratory Distress Syndrome.
9. To compare and validate different risk scores in our cohort.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years old admitted to ICU with Severe Septic Shock

Exclusion Criteria:

* Rejecting participation by not signing informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe Septic Shock defined by requiring norepinephrine at more than 0.25mcg/kg/min
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Lactate clearance | 30 days
  Time from hospital arrival to documented serum lactate of less than or equal to 2 mmol/L

SECONDARY OUTCOMES:
Days alive and free of Mechanical Ventilation, Vasopressors and Renal Replacement Therapy | 28 days
  Number of days from the last day free of vasopressors, mechanical ventilation and Renal Replacement Therapy up to day 28. If patients dies it scores 0.
Mechanical Ventilation-free days | 28 days
  Days free of mechanical ventilation up to day 28
Vasopressors-free days | 28 days
  Days free of vasopressors up to day 28
Rate of Acute Kidney Injury | 28 days
  Kidney Disease: Improving Global Outcomes definition
ICU length of stay | 28 days
  Days in ICU
Hospital length of stay | 30 days
  Days in Hospital
Rate of In-hospital Mortality | 30 days
  Any cause mortality
Rate of Acute Respiratory Distress Syndrome | 28 days
  Berlin definition
Rate of New Atrial Fibrilation | 28 days
  New atrial fibrilation requiring treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Venot M, Weis L, Clec'h C, Darmon M, Allaouchiche B, Goldgran-Toledano D, Garrouste-Orgeas M, Adrie C, Timsit JF, Azoulay E. Acute Kidney Injury in Severe Sepsis and Septic Shock in Patients with and without Diabetes Mellitus: A Multicenter Study. PLoS One. 2015 May 28;10(5):e0127411. doi: 10.1371/journal.pone.0127411. eCollection 2015. PMID 26020231
- [Background] Barbar SD, Clere-Jehl R, Bourredjem A, Hernu R, Montini F, Bruyere R, Lebert C, Bohe J, Badie J, Eraldi JP, Rigaud JP, Levy B, Siami S, Louis G, Bouadma L, Constantin JM, Mercier E, Klouche K, du Cheyron D, Piton G, Annane D, Jaber S, van der Linden T, Blasco G, Mira JP, Schwebel C, Chimot L, Guiot P, Nay MA, Meziani F, Helms J, Roger C, Louart B, Trusson R, Dargent A, Binquet C, Quenot JP; IDEAL-ICU Trial Investigators and the CRICS TRIGGERSEP Network. Timing of Renal-Replacement Therapy in Patients with Acute Kidney Injury and Sepsis. N Engl J Med. 2018 Oct 11;379(15):1431-1442. doi: 10.1056/NEJMoa1803213. PMID 30304656
- [Background] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185
- [Background] McIntyre WF, Um KJ, Alhazzani W, Lengyel AP, Hajjar L, Gordon AC, Lamontagne F, Healey JS, Whitlock RP, Belley-Cote EP. Association of Vasopressin Plus Catecholamine Vasopressors vs Catecholamines Alone With Atrial Fibrillation in Patients With Distributive Shock: A Systematic Review and Meta-analysis. JAMA. 2018 May 8;319(18):1889-1900. doi: 10.1001/jama.2018.4528. PMID 29801010